CLINICAL TRIAL: NCT04331834
Title: Pre-Exposure Prophylaxis With Hydroxychloroquine for High-Risk Healthcare Workers During the COVID-19 Pandemic: A Multicentre, Double-Blinded Randomized Controlled Trial
Brief Title: Pre-Exposure Prophylaxis With Hydroxychloroquine for High-Risk Healthcare Workers During the COVID-19 Pandemic
Acronym: PrEP_COVID
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Barcelona Institute for Global Health (Other)
Collaborators: Hospital Clinic of Barcelona (Other); Laboratorios Rubió (Unknown); Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other); Hospital Plató (Other); Hospital de Granollers (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PrEP_COVID
Record Dates: First submitted 2020-04-01; First posted 2020-04-02 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: COVID-19
Keywords: PrEP; hydroxychloroquine; prophylaxis; pre-exposure; healthcare workers
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pre-exposure prophylaxis of SARS-CoV-2 (Experimental): Participants will receive hydroxychloroquine 400 mg daily during the first 4 days, followed by 400 mg weekly during 6 months
  Interventions: Drug: Hydroxychloroquine
- Control group with placebo (Placebo Comparator): Participants will receive placebo 400 mg daily during the first 4 days, followed by 400 mg weekly during 6 months
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Hydroxychloroquine — Hydroxychloroquine with the following dosage:
  * day 0: 400 mg (2 tablets)
  * day 1: 400 mg (2 tablets)
  * day 2: 400 mg (2 tablets)
  * day 3: 400 mg (2 tablets)
  * weekly: 400 mg (2 tablets) for a period of six months
  Arms: Pre-exposure prophylaxis of SARS-CoV-2
Drug: Placebos — Placebo with the following dosage:
  * day 0: 400 mg (2 tablets)
  * day 1: 400 mg (2 tablets)
  * day 2: 400 mg (2 tablets)
  * day 3: 400 mg (2 tablets)
  * weekly: 400 mg (2 tablets) for a period of six months
  Arms: Control group with placebo

SUMMARY:
The investigators aim to evaluate the efficacy of pre-exposure prophylaxis with hydroxychloroquine in healthcare workers with high-risk of SARS-CoV-2 infection.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Negative PCR and negative serology on day 0
* Healthcare worker at any of the trial sites
* Female participants: negative for pregnancy test
* Willing to participate in the study
* Able to sign the informed consent form

Exclusion Criteria:

* Age <18 years
* Pregnancy or breastfeeding
* Ongoing antiviral or antiretroviral treatment or HIV positive
* Ongoing anti-inflammatory treatment (corticosteroids)
* Ongoing or previous (1 month) chloroquine or hydroxychloroquine treatment
* Confirmed case of SARS-CoV-2 infection (positive PCR) at day 0
* Positive serology for SARS-CoV-1 infection at day 0
* Impossibility of signing the informed consent form
* Rejection of participation
* Working less than 3 days a week in the Hospital Clinic of Barcelona.
* Any contraindication for hydroxychloroquine treatment:

  * Hydroxychloroquine hypersensitivity or 4-aminoquinoline hypersensitivity
  * Retinopathy, visual field or visual acuity disturbances
  * QT prolongation, bradycardia (<50bpm), ventricular tachycardia, other arrhythmias, as determined on day 0 ECG or medical history
  * Potassium < 3 mEq/L or AST or ALT > 5 upper normal limit, as determined on day 0 blood test
  * Previous myocardial infarction
  * Myasthenia gravis
  * Porphyria
  * Glomerular clearance < 10ml/min
  * Previous history of severe hypoglycaemia
  * Ongoing treatment with antimalarials, antiarrhythmic, tricyclic antidepressants, selective serotonin reuptake inhibitors, natalizumab, quinolones, macrolides, agalsidase alfa and beta.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2020-04-03 (Actual); Primary Completion 2020-06-25 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Confirmed cases of a COVID-19 | Up to 6 months after start of treatment
  Confirmed cases of a COVID-19 (defined by a positive PCR for SARS-CoV-2 or symptoms compatible with COVID-19 with seroconversion) in the PrEP group compared to the placebo group at any time during the 6 months of the follow-up in healthcare workers with negative PCR for SARS-CoV-2 on day 0 and negative serology for SARS-CoV-2 on day 0.

SECONDARY OUTCOMES:
SARS-CoV-2 seroconversion | Up to 6 months after start of treatment
  SARS-CoV-2 seroconversion in the PrEP group compared to placebo in during 6 months of follow-up in healthcare workers with negative serology at day 0.
Occurrence of any adverse event related with hydroxychloroquine treatment | Up to 6 months after start of treatment
  Incidence of clinical and/or laboratory adverse events will be compared in the PrEP group and in the placebo arm.
Incidence of SARS-CoV-2 infection and COVID-19 among healthcare workers | Up to 6 months after start of treatment
  Incidence of SARS-CoV-2 infection and COVID-19 among healthcare workers will be estimated by the number of healthcare workers diagnosed with COVID-19 in the placebo group, among the total of healthcare workers included in the non-PrEP group during the study period.
Risk ratio for the different clinical, analytical and microbiological conditions to develop COVID-19 | Up to 6 months after start of treatment
COVID-19 Biobank | Up to 6 months after start of treatment
  A repository (biobank) of serum samples obtained from healthcare workers confirmed COVID-19 cases for future research on blood markers to predict SARS-CoV-2 infection.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Muñoz Gutiérrez, MD, PhD, Principal Investigator — Barcelona Institute for Global Health
Locations (1):
- ISGlobal, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grau-Pujol B, Camprubi-Ferrer D, Marti-Soler H, Fernandez-Pardos M, Carreras-Abad C, Andres MV, Ferrer E, Muelas-Fernandez M, Jullien S, Barilaro G, Ajanovic S, Vera I, Moreno L, Gonzalez-Redondo E, Cortes-Serra N, Roldan M, Arcos AA, Mur I, Domingo P, Garcia F, Guinovart C, Munoz J. Pre-exposure prophylaxis with hydroxychloroquine for COVID-19: a double-blind, placebo-controlled randomized clinical trial. Trials. 2021 Nov 15;22(1):808. doi: 10.1186/s13063-021-05758-9. PMID 34781981
- [Derived] Grau-Pujol B, Camprubi D, Marti-Soler H, Fernandez-Pardos M, Guinovart C, Munoz J. Pre-exposure prophylaxis with hydroxychloroquine for high-risk healthcare workers during the COVID-19 pandemic: A structured summary of a study protocol for a multicentre, double-blind randomized controlled trial. Trials. 2020 Jul 29;21(1):688. doi: 10.1186/s13063-020-04621-7. PMID 32727613